CLINICAL TRIAL: NCT02498574
Title: Performance Enhancement and Non-Invasive Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: M16-15-015
Record Dates: First submitted 2015-07-09; First posted 2015-07-15 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Executive Function; Motor Activity; Brain Stimulation
MeSH Terms: conditions — Motor Activity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Group 1 (Experimental): Non-invasive brain stimulation protocol expected to improve performance, with cognitively challenging game
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Working Memory Training
- Group 2 (Placebo Comparator): Non-invasive brain stimulation protocol not expected to improve performance, with cognitively challenging game
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Working Memory Training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Non-invasive brain stimulation applied to the surface of the scalp
Behavioral: Working Memory Training — Cognitively challenging game played concurrently with transcranial direct-current stimulation

SUMMARY:
A promising form of enhancing brain function non-invasively involves stimulating the brain using weak magnetic or electric currents. This method is becoming increasingly popular in both clinical and commercial circles; a number of portable, at-home devices are available on the commercial market for personal use. In this study, the investigators aim to determine factors associated with the enhancement of cognitive and motor learning following transcranial direct-current stimulation in healthy young adults. Understanding how participants respond to brain stimulation is critical to maximizing the effectiveness of stimulation and determining its potential as a performance-enhancing aid for mental tasks. Future developments of this study may also inform the capacity of brain stimulation to act as non-drug alternative to treatment for cognitive decline.

DETAILED DESCRIPTION:
This study involves a single session of anodal tDCS, applied over the motor cortex, while performing a task of motor dexterity. Pre and post stimulation evaluations will assess any effects of the stimulation on motor and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in good health,
* between 18-35 years of age
* with no prior history of neurological diseases such as multiple sclerosis, Parkinson's disease, stroke with paralysis.

Exclusion Criteria:

* Participants with cardiac stimulators (pace-makers) and those with metal implants in the skull will be excluded.
* Pregnant women will also be excluded.

Participants will be required to fill out a brief health questionnaire to ensure that they have no conditions that would prevent brain stimulation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in ratings on cognitive training survey | Baseline, Post-test following 20-minute stimulation period
  This survey aims to assess participant perceptions on brain stimulation, and includes a series of related questions, rated on a scale of 1-7.
Change in cognitive performance | Baseline, Post-test following 20-minute stimulation period
  We will measure changes in cognitive performance on neuropsychological tests.
Change in game performance | Baseline, Post-test following 20-minute stimulation period
  We will measure changes in performance on a cognitively-challenging game performed concurrently with the non-invasive brain stimulation.
Change in motor performance | Baseline, Post-test following 20-minute stimulation period
  We will measure changes in motor performance on the Grooved Pegboard task.

CONTACTS AND LOCATIONS:
Overall Officials: Sheida Rabipour, PhD, Principal Investigator — University of Ottawa; Francois Tremblay, PT, PhD, Principal Investigator — Bruyere Continuing Care; Patrick SR Davidson, PhD, Principal Investigator — University of Ottawa
Locations (2):
- Canada (2):
  - Bruyere Continuing Care, Ottawa, Ontario
  - Bruyere Research Institute, Ottawa, Ontario